CLINICAL TRIAL: NCT07088380
Title: The Additive Effect of Ketamine in Combination With ElectroConvulsive Stimulation (ECS) in Major Depressive Disorder (MDD): a Translational Study
Brief Title: Ketamine Augmentation of ECT in Treatment-Resistant Depression
Acronym: Ketamina
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Full Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRIN - 20227EA9AN
Record Dates: First submitted 2025-07-08; First posted 2025-07-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
Keywords: ketamine; TRD; depression; electroconvulsive therapy (ECT)
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Patients receive standard ECT treatment combined with intravenous ketamine at a subanesthetic dose of 0.5 mg/kg, administered after induction with Propofol. Ketamine is administered during ECT sessions 2, 4, and 6.
  Intervention:
  * Drug: Ketamine
  * Dose: 0.5 mg/kg IV
  * Timing: ECT sessions 2, 4, and 6
  * Background: Investigating the additive antidepressant and potential cognitive-protective effects of ketamine in patients with treatment-resistant depression undergoing ECT.
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): Patients receive standard ECT treatment combined with placebo (0.9% sodium chloride solution), administered intravenously after induction with Propofol, during ECT sessions 2, 4, and 6, mimicking the ketamine group's schedule.
  Intervention:
  * Drug: Saline solution (NaCl 0.9%)
  * Timing: ECT sessions 2, 4, and 6
  * Background: Serves as control to assess the specific contribution of ketamine to antidepressant efficacy and cognitive outcomes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine will be administered intravenously at a subanesthetic dose of 0.5 mg/kg after a bolus of Propofol, during ECT sessions 2, 4, and 6.
  Arms: Ketamine
Drug: Placebo — Placebo will be administered intravenously at a subanesthetic dose of 0.5 mg/kg after a bolus of Propofol, during ECT sessions 2, 4, and 6.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 3 clinical trial evaluating the additive effect of intravenous ketamine in combination with electroconvulsive therapy (ECT) in patients with treatment-resistant major depressive disorder (MDD). The study aims to determine whether ketamine enhances the antidepressant efficacy of ECT and reduces associated cognitive side effects. Thirty hospitalized patients diagnosed with treatment-resistant MDD will be randomized to receive either ketamine or placebo (saline) during ECT sessions 2, 4, and 6. Primary outcome is the change in depressive symptoms, measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18-70,
* diagnosed with MDD (according to SCID5-CV interview)
* treatment resistant (defined as at least 2 different antidepressant agents used without success),
* ability to give informed consent,
* adequacy of the score for anesthesia.

Exclusion Criteria:

* Chronic neurological diseases,
* Intellectual disability
* Contraindications to the electroconvulsive therapy (severe aortic valve stenosis, implantable cardiac defibrillators, uncontrolled hypertension, clinically significant respiratory, renal or hepatic disease, abdominal aortic aneurysm, endocrine disorders, neuromuscular diseases, space occupying brain lesions, stroke in the last 6 months),
* Patients with Alcohol Use Disorder or Substance Use Disorder or Substance Abuse history in the past year,
* Pregnancy and lactation
* Cardiovascular conditions,
* Psychiatric Disorders,
* Hepatic impairment,
* Participants with a known hypersensitivity to ketamine or any of its excipients will be excluded from the study,
* Participants with any contraindications to the use of ketamine, such as a history of severe cardiovascular conditions (e.g., uncontrolled hypertension, significant arrhythmias), intracranial hypertension, or severe liver impairment, will also be excluded to prevent potential adverse events.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Mean change in depressive symptoms, as measured by MADRS scale | From baseline (day 0) to day 28 (7 days after the last ECT session). A follow-up assessment at Week 12 (90 days) will be included
  The primary efficacy endpoint will be assessed using the MADRS score (Montgomery-Åsberg Depression Rating Scale)

SECONDARY OUTCOMES:
Change in Suicidal Ideation (Beck Scale for Suicide Ideation - BSSI) | Assessment will be performed at: baseline (day 0); Weekly during ECT treatment period (Weeks 1, 2, 3); Week 4 (1 week after last ECT session); Follow-up: Week 12 (3 months after last ECT session)
  To assess the effect of ketamine and ECT on suicidal ideation with Beck Scale for Suicide Ideation (BSSI)
Change in Anxiety Symptoms (Hamilton Anxiety Rating Scale - HAM-A) | Assessment will be performed at: baseline (day 0); Weekly during ECT treatment period (Weeks 1, 2, 3); Week 4 (1 week after last ECT session); Follow-up: Week 12 (3 months after last ECT session)
  To evaluate the impact of ketamine and ECT on anxiety symptoms with Hamilton Anxiety Rating Scale (HAM-A)
Change in Cognitive Function (Brief Assessment of Cognition in Affective Disorders - BAC-A) | Assessment will be performed at: baseline (day 0); Week 4 (1 week after last ECT session); Follow-up: Week 12 (3 months after last ECT session)
  To determine the cognitive effects of ketamine and ECT with Brief Assessment of Cognition in Affective Disorders (BAC-A)
Change in Dissociative and Psychotic Symptoms (Clinician-Administered Dissociative States Scale - CADSS; Brief Psychiatric Rating Scale - BPRS) | Assessment will be performed at: Baseline (Day 0, before first ECT session); Week 1 (After ECT session 2); Week 2 (After ECT session 4); Week 3 (After ECT session 6); Week 4 (1 week after last ECT session); Follow-up: Week 12 (3 months after last ECT
  To assess the effects of ketamine and ECT on dissociative and psychotic symptoms with Clinician-Administered Dissociative States Scale (CADSS) and Brief Psychiatric Rating Scale (BPRS)
Change in Neurochemical Markers (Plasma Levels of Trp, 5-HT, 5-HIAA, Glutamate, Aspartate) | Assessment will be performed at: Baseline (Day 0, before first ECT session); Weekly during ECT treatment period (Weeks 1, 2, 3)
  To evaluate the neurochemical effects of ketamine and ECT with High-Performance Liquid Chromatography (HPLC) analysis of plasma samples. Change in plasma levels of Trp, 5-HT, 5-HIAA, glutamate, and aspartate from baseline to Week 3 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto AZ Zangrillo, MD, Principal Investigator — Università Vita-Salute San Raffaele; Cristina CC Colombo, MD, Principal Investigator — IRCCS Ospedale San Raffaele Turro
Locations (1):
- IRCCS Ospedale San Raffaele Turro, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz J, Murrough JW, Iosifescu DV. Ketamine for treatment-resistant depression: recent developments and clinical applications. Evid Based Ment Health. 2016 May;19(2):35-8. doi: 10.1136/eb-2016-102355. Epub 2016 Apr 6. PMID 27053196
- [Background] Anderson IM, Blamire A, Branton T, Clark R, Downey D, Dunn G, Easton A, Elliott R, Elwell C, Hayden K, Holland F, Karim S, Loo C, Lowe J, Nair R, Oakley T, Prakash A, Sharma PK, Williams SR, McAllister-Williams RH; Ketamine-ECT Study team. Ketamine augmentation of electroconvulsive therapy to improve neuropsychological and clinical outcomes in depression (Ketamine-ECT): a multicentre, double-blind, randomised, parallel-group, superiority trial. Lancet Psychiatry. 2017 May;4(5):365-377. doi: 10.1016/S2215-0366(17)30077-9. Epub 2017 Mar 27. PMID 28359862
- [Background] Fava M, Freeman MP, Flynn M, Judge H, Hoeppner BB, Cusin C, Ionescu DF, Mathew SJ, Chang LC, Iosifescu DV, Murrough J, Debattista C, Schatzberg AF, Trivedi MH, Jha MK, Sanacora G, Wilkinson ST, Papakostas GI. Double-blind, placebo-controlled, dose-ranging trial of intravenous ketamine as adjunctive therapy in treatment-resistant depression (TRD). Mol Psychiatry. 2020 Jul;25(7):1592-1603. doi: 10.1038/s41380-018-0256-5. Epub 2018 Oct 3. PMID 30283029
- [Background] Nuzzi M, Delmonte D, Barbini B, Pasin L, Sottocorna O, Casiraghi GM, Colombo C, Landoni G, Zangrillo A. Thiopental is better than propofol for electroconvulsive therapy. Acta Biomed. 2018 Jan 16;88(4):450-456. doi: 10.23750/abm.v88i4.6094. PMID 29350659